CLINICAL TRIAL: NCT04910555
Title: Is Strong Desire to Void an Equivalent of Cognitive Task Affecting Balance in Older Women With Overactive Bladder?
Brief Title: Strong Desire to Void and Balance in Older Women With Overactive Bladder
Acronym: SURFACE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210072; 2021-A00406-35 (Other: IDRCB Number)
Record Dates: First submitted 2021-04-29; First posted 2021-06-02 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Overactive Bladder; Urinary Incontinence
Keywords: balance; strong desire to void; older women; overactive bladder; cognitive task
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women over 65 years old with OAB: Community-dwelling women over 65 years old, with non-neurogenic OAB, with or without UI
  Interventions: Other: strong desire to void - cognitive task

INTERVENTIONS:
Other: strong desire to void - cognitive task — Strong desire to void - cognitive task (verbal fluency)

SUMMARY:
Falls have multifactorial etiologies in older people. Lower urinary tract symptoms (LUTS) are one of those, with an increase prevalence over years (30% of people over 75 years old have overactive bladder [OAB]). Previous studies showed that older women with OAB with or without urinary incontinence (UI) are prone to have gait disorders (decrease of gait speed and step width and increase of number of step). Besides UI, it is more likely the strong desire to void (SDV) that seems to impact gait and balance control. In older women with UI, balance on stabilometric parameters have been affected with an increase of the center of pression (COP) sway range, COP area and rambling trajectory. SDV seems to act like an additional cognitive task. A similar and increased reaction time has been observed in comparing with a distracting task in healthy volunteers. In older people who are susceptible to distracting task, SDV may alters balance and gait.

The primary objective of this prospective study is to assess the impact of SDV on stabilometric parameters (center of foot pressure (COP) area, the distance travelled made by COP, the mean X-axis displacement and the mean Y-axis displacement) compared to the "empty bladder" condition.

The secondary objectives are to assess the impact of a cognitive task (verbal fluency) on stabilometric parameters in comparison with the "no cognitive task condition" and the "SDV condition"; to assess the impact of "SDV condition" on balance and gait clinical evaluation (Timed up and go test, unipedal stance test, Berg scale, 10m walking speed, 5 chair stand) Thus, showing that SDV may impact balance in geriatric population will lead to the importance to identify and LUTS as potential fall risk factor in order to decrease falls incidence in this population.

DETAILED DESCRIPTION:
Falls have multifactorial etiologies in older people. Lower urinary tract symptoms (LUTS) are one of those, with an increase prevalence over years (30% of people over 75 years old have overactive bladder [OAB]). Previous studies showed that older women with oAB with or without urinary incontinence (UI) are prone to have gait disorders (decrease of gait speed and step width and increase of number of step). Besides UI, it is more likely the strong desire to void (SDV) that seems to impact gait and balance control. In older women with UI, balance on stabilometric parameters has been affected with an increase of the center of pression (COP) sway range, COP area and rambling trajectory. SDV seems to act like an additional cognitive task.

A similar and increased reaction time has been observed in comparing with a distracting task in healthy volunteers. In older people who are susceptible to distracting task, SDV may alters balance and gait.

The primary objective of this prospective study is to assess the impact of SDV on stabilometric parameters (center of foot pressure (COP) area, the distance travelled made by COP, the mean X-axis displacement and the mean Y-axis displacement) compared to the "empty bladder" condition.

The secondary objectives are assessing the impact of a cognitive task (verbal fluency) on stabilometric parameters in comparison with the "no cognitive task condition" and the "SDV condition"; and assessing the impact of "SDV condition" on balance and gait clinical evaluation (Timed up and go test, unipedal stance test, Berg scale, 10m walking speed, 5 chair stand) This prospective study will take place in a rehabilitation department during a 2hours-consultation. The eligible criteria are: women over 65 years old, with OAB with or without UI, able to walk without mobility equipment without neurologic pathology or spine surgery, without severe cognitive impairment (MMSE > 24) or legal protection, and who agree to be involved in the study. OAB was defined by urinary urgency, usually with urinary frequency and nocturia, with or without urgency urinary incontinence.

The included women will first have a standard urinary consultation in which comorbidities, treatments and urinary symptoms will be recorded. Participants will also have questionnaires on urinary symptoms (Urinary Symptom Profile and Incontinence Consultation Incontinence Questionnaires) and the Mini Mental Status Examination (assessing cognitive functions).

Then, participants will be evaluated on balance and gait clinical and instrumental parameters under "SDV" and "empty bladder" conditions. The order of these evaluations (SDV/empty bladder) is randomized by computer. The clinical evaluations are the Timed up and go test, the unipedal stance test, the Berg scale, the 10m walking speed test and the 5-chair-stand test. The stabilometry evaluation (recording the center of foot pressure (COP) area, the distance travelled made by COP, the mean X-axis displacement and the mean Y-axis displacement) will be on a force platform under 4 conditions: SDV with and without verbal fluency and empty bladder with and without verbal fluency.

The stabilographic parameters will be analyzed using a two-way repeated measures ANOVAs. The repeated factors are the SDV and empty bladder condition and with or without verbal fluency. Four testing combinations of these factors will be used: SDV/with verbal fluency, SDV/without verbal fluency, empty bladder/with verbal fluency and empty bladder/without verbal fluency. The ANOVA results will be used to calculate the F statistics for each main effect and interaction. The post-hoc comparisons will be performed using the Bonferroni test. The level of statistical significance was set in all tests at P≤0.05.

Thus, if we show that SDV may impact balance in geriatric population it will lead to the importance to identify and treat LUTS as potential fall risk factor in order to decrease falls incidence in this population.

ELIGIBILITY:
Inclusion Criteria:

* women;
* over 65 years old;
* with OAB with or without UI;
* able to walk without mobility aid; consent to participate in the study

Exclusion Criteria:

* neurologic pathology; history of spine surgery;
* cognitive impairment defined as a MMSE < 24;
* legal protection

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Community-dweeling women over 65 years old, with non-neurogenic OAB, with or without UI
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Stabilometry platform assesment | 1 day
  The primary outcome is a composite criterion of 4 parameters, assessing changes in stabilometry platform between "strong desire to void" and "empty bladder" conditions. These 4 parameters are the center of foot pressure (COP) area, the distance travelled made by COP, the mean X-axis displacement and the mean Y-axis displacement. need for bladder emptiness).

SECONDARY OUTCOMES:
Clinical balance | 1 day
  Comparison of the Timed up and go test results between the 2 conditions: "strong desire to void" and "empty bladder".
Gait assesment | 1 day
  Gait assesment: 10m walking speed
cognitive task assesment | 1 day
  cognitive task evaluation ( words per minute) during B3 compared to B0 ( absence of need for bladder emptiness).bladder" conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No